CLINICAL TRIAL: NCT00047190
Title: A Phase II Trial of R115777 in Myelofibrosis With Myeloid Metaplasia (MMM)
Brief Title: Tipifarnib in Treating Patients With Myelofibrosis and Myeloid Metaplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02804; MC0184; N01CM17104 (NIH)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera; Primary Myelofibrosis
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — tipifarnib

ARMS (1):
- Arm I (Experimental): Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of tipifarnib in treating patients who have myelofibrosis with myeloid metaplasia. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate in MMM patients treated with R115777. II. To evaluate the toxicity of R115777 in patients with MMM.

SECONDARY OBJECTIVES:

I. To evaluate the benefit of therapy with R115777 in alleviating disease-associated anemia in patients with MMM.

II. To evaluate the benefit of R115777 in reducing palpable splenomegaly in patients with MMM.

III. To evaluate the effect of R115777 on the hypercatabolic symptoms from MMM. IV. To evaluate the effect of R115777 on the pathologic increase in circulating myeloid progenitors in MMM patients through baseline measurement and measurement after the first cycle.

V. To correlate response/relapse with in vitro myeloid colony sensitivity to R115777 at the time of either response or relapse.

VI. To evaluate the effect of R115777 on bone marrow histologic features of MMM including osteosclerosis, reticulin fibrosis, and angiogenesis (through serial bone marrow microvessel density grading).

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 2 years.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study within 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmation (on bone marrow trephine and aspirate) of myelofibrosis with myeloid metaplasia by a pathologist/hematologist at the registering institution; included in the diagnosis of MMM are AMM (agnogenic myeloid metaplasia), PPMM (post-polycythemic myeloid metaplasia), and PTMM (post-thrombocythemic myeloid metaplasia); the bone marrow should show the presence of reticulin fibrosis, and the peripheral blood smear should show the presence of leukoerythroblastosis and dacrocytosis
* Bone marrow showing no evidence of other conditions associated with myelofibrosis, such as metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease, acute leukemia (including M7 type), or acute myelofibrosis
* Bone marrow chromosome analysis or peripheral blood or bone marrow Fluorescent In Situ Hybridization (FISH) showing absence of chromosomal translocation t(9:22); prior demonstration is sufficient for enrollment purposes
* At least one of the following:

  * Anemia evidenced by hemoglobin < 10 g/dL
  * Palpable hepato-splenomegaly
* ANC ≥ 750/mm^3
* PLT ≥ 100,000/mm^3
* Total bilirubin (direct if total elevated) ≤ UNL
* Alkaline phosphatase =< 3 x UNL (unless felt to be secondary to disease)
* AST ≤ 2.5 x UNL
* Creatinine =< 1.5 x UNL
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to follow the schedule for returning to the registering P2C institution (monthly) while receiving protocol treatment
* ECOG performance status 0, 1, or 2

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
  * NOTE: The effects of the agent(s) on the developing human fetus at the recommended therapeutic dose are unknown
* Use of cytotoxic chemotherapy or other myelosuppressive agents within =< 2 weeks prior to study entry
* Uncontrolled intercurrent illness or any co-morbid condition that would limit compliance with study requirements or with which the use of R115777 is felt to be potentially harmful; such conditions include, but are not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia, or
  * Psychiatric illness/social situations
* Other concurrent therapy directed at the disease (including Thalidomide) or use of erythropoietin while enrolled in this study; such agents must be discontinued at the time of or prior to study entry
* Known quinolone sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Confirmed response defined as the objective status of complete response (CR) or partial response (PR) on 2 consecutive evaluations at least 4 weeks apart | Up to 2 years
  Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall survival | Time from registration to death due to any cause, assessed up to 2 years
  Estimated using the method of Kaplan-Meier.
Time to progression | Time from registration to the time of progression, assessed up to 2 years
  Estimated using the method of Kaplan-Meier.
Duration of response | Date of complete response to the date progression is documented (if one has occurred) or to the date of last follow-up (for those patients who have not progressed), assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Mesa, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States